CLINICAL TRIAL: NCT07270848
Title: A Multicenter Prospective Study on the Efficacy, Safety, and Quality of Life Improvements of Dronedarone for Early Rhythm Control in Atrial Fibrillation
Brief Title: Dronedarone Rhythm Intervention for Early Atrial Fibrillation
Acronym: DRIVE-AF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Yong-Soo Baek, Associate Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-06-013
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Dronedarone; Flecainide; Propafenone; Antiarrhythmic Drugs; Rhythm Control
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone; Unmanned Aerial Devices; Flecainide; Propafenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronedarone (Experimental): Participants assigned to this arm will receive dronedarone 400 mg twice daily.
  Interventions: Drug: Dronedarone
- Class Ic Antiarrhythmic Drugs (Active Comparator): Participants assigned to this arm will receive a Class Ic antiarrhythmic drug (investigator's choice of flecainide or propafenone) according to standard clinical practice.
  Interventions: Drug: flecainide; Drug: propafenone

INTERVENTIONS:
Drug: Dronedarone — Dronedarone 400 mg administered orally twice daily.
  Other Names: Multaq; Drone Tab.
  Arms: Dronedarone
Drug: flecainide — Administered orally according to standard clinical practice.
  Other Names: Tambocor
  Arms: Class Ic Antiarrhythmic Drugs
Drug: propafenone — Administered orally according to standard clinical practice.
  Other Names: Rytmonorm
  Arms: Class Ic Antiarrhythmic Drugs

SUMMARY:
The purpose of this study is to compare two commonly used types of medicine for treating atrial fibrillation (also called AF), a condition that causes an irregular heart rhythm. This study is for adults who have been diagnosed with AF within the past year.

Researchers want to find out which medicine is more effective, safer, and provides a better quality of life for patients needing to control their heart rhythm.

Participants who agree to join the study will be randomly assigned (like flipping a coin) to one of two groups:

Group 1: Will receive the medicine Dronedarone.

Group 2: Will receive a standard medicine from the 'Class Ic' group (such as flecainide or propafenone).

The study will follow participants for at least 12 months. Researchers will compare how well each medicine works to prevent AF from coming back. They will also carefully track any side effects and changes in participants' quality of life during the study.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, open-label trial designed to address a common clinical question in the management of recent-onset atrial fibrillation (AF). Following recent evidence supporting the benefits of an early rhythm-control strategy, both dronedarone and Class Ic antiarrhythmic drugs (AADs) are widely used. However, there is a lack of large-scale, prospective, randomized data directly comparing the efficacy, safety, and quality of life outcomes between these two treatment strategies in this specific population.

The primary objective of the DRIVE-AF study is to compare the clinical outcomes of dronedarone versus standard Class Ic AADs (flecainide or propafenone) in patients with AF diagnosed within the past year.

Approximately 1,898 participants will be enrolled at 16 centers in the Republic of Korea. Eligible participants who provide informed consent will be randomized in a 1:1 ratio to receive either dronedarone or a Class Ic AAD (investigator's choice of flecainide or propafenone).

All participants will be followed for a minimum of 12 months. Efficacy will be primarily assessed by the recurrence of atrial fibrillation. Safety endpoints, particularly the rate of drug discontinuation due to adverse events, and patient-reported outcomes, including quality of life measured by the AF-QoL questionnaire, will be systematically collected and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have voluntarily provided written informed consent to participate.
* Adults aged 19 years or older.
* Life expectancy of at least 1 year.
* Diagnosis of atrial fibrillation within the past 1 year.
* Participants with an indication for antiarrhythmic drug therapy (Dronedarone or Class Ic agents).

Exclusion Criteria:

* History of failure with prior antiarrhythmic drug therapy.
* Confirmed severe structural heart disease (e.g., heart failure with reduced ejection fraction [LVEF <= 40%], moderate or severe mitral stenosis, mechanical heart valve replacement, or dilated cardiomyopathy).
* Diagnosis of permanent atrial fibrillation.
* Severe renal impairment (eGFR < 30 mL/min/1.73m^2 or on dialysis) or severe hepatic impairment (Child-Pugh class B or higher) that restricts the use of antiarrhythmic drugs.
* Known contraindications to dronedarone or Class Ic antiarrhythmic drugs.
* Participation in another clinical trial within 3 months prior to randomization.
* Participants who do not agree to refrain from participating in another clinical trial within 14 days after their participation in this study ends.
* Pregnant or breastfeeding women, or women of childbearing potential who do not agree to use effective contraception during the study.
* Any other condition that, in the opinion of the investigator, makes the participant unsuitable for study participation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1898 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy : Recurrence of Atrial Fibrillation | From randomization up to 12 months
  Percentage of participants who experience a recurrence of atrial fibrillation (AF), atrial flutter, or atrial tachycardia lasting 30 seconds or more, as documented by 12-lead ECG, 24-hour Holter monitoring or wearable Holter monitoring
Safety : Rate of Drug Discontinuation Due to Adverse Events | Up to 12 months
  Percentage of participants who permanently discontinue the assigned study drug due to any adverse event (AE) or serious adverse event (SAE).

SECONDARY OUTCOMES:
Change in Atrial Fibrillation-Specific Quality of Life (AF-QoL) | The change in scores will be compared between enrollment (baseline) and the 12-month time point.
  The impact of early rhythm control on quality of life will be assessed using the Atrial Fibrillation Quality of Life (AF-QoL) questionnaire. This questionnaire includes items related to psychological, physical, and sexual activity. The total score is standardized to a scale ranging from 0 to 100, with higher scores indicating a better quality of life.
Medication Adherence | 6 months and 12 months
  The proportion of patients who remain on the assigned study medication will be measured. Adherence will be assessed using the Proportion of Days Covered (PDC) calculation. A PDC of 80% or greater is defined as adherent.
Comparison of Atrial Fibrillation Treatment Options | Up to 12 months
  To assess the rates of: (a) use of Non-vitamin K Antagonist Oral Anticoagulants (NOACs), (b) use of medical therapy (rate control and rhythm control), (c) atrial fibrillation catheter ablation, and (d) direct current cardioversion (DCCV).
Incidence of Other Arrhythmias on Holter or Wearable Patch ECG | Up to 12 months
  To compare the detection rate of other arrhythmias (e.g., Premature Atrial Contractions (PAC), Premature Ventricular Contractions (PVC), Atrioventricular (AV) Block, Supraventricular Tachycardia (SVT), and Ventricular Tachycardia (VT)) documented by Holter or wearable patch ECG monitoring.
Incidence of Major Adverse Cardiovascular Events (MACE) | Up to 12 months
  To measure the incidence of: (a) cardiovascular death, (b) stroke, (c) hospitalization for worsening heart failure, and (d) hospitalization for acute coronary syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Soo Baek, M.D., Ph.D., Study Chair — Division of Cardiology, Department of Internal Medicine, Inha University College of Medicine and Inha University Hospital, Incheon, Republic of Korea.
Locations (16):
- South Korea (16):
  - Inha University Hospital, Incheon, Incheon
  - Korea University Ansan Hospital, Ansan
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Kosin University Gospel Hospital, Busan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Inje University Ilsan Paik Hospital, Goyang
  - NHIS Ilsan Hospital, Goyang-si
  - Myongji Hospital, Goyang-si
  - Hanyang University Guri Hospital, Guri-si
  - Jeju National University Hospital, Jeju City
  - Sejong Chungnam National University Hospital, Sejong
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect the privacy of study participants. The informed consent form signed by the participants does not include a provision for data sharing with third parties.